CLINICAL TRIAL: NCT01472965
Title: A Double-Blind, Randomized, Placebo-Controlled, Trial of Ethanol Lock Therapy for Treatment and Secondary Prophylaxis of Central Line Associated Bloodstream Infection (CLABSI) in Children and Adolescents
Brief Title: Ethanol Lock Therapy for Treatment and Secondary Prophylaxis of Central Line-Associated Bloodstream Infection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ETHEL
Record Dates: First submitted 2011-11-14; First posted 2011-11-17 (Estimated); Results first posted 2017-11-13 (Actual); Last update posted 2017-11-13 (Actual); Status verified 2017-08

CONDITIONS: Central Line-Associated Bloodstream Infection
Keywords: central line; adolescents; children; bloodstream infection; antibiotic lock therapy; catheter lock therapy; ethanol lock therapy
MeSH Terms: conditions — Sepsis | interventions — Ethanol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment (Active Comparator): Eligible patients with CLABSI will be enrolled within 96 hours of collection of positive blood culture and randomized to blinded treatment with 70% ethanol catheter lock therapy.
  Interventions: Drug: ethanol
- Control (Placebo Comparator): Eligible patients with CLABSI will be enrolled within 96 hours of collection of positive blood culture and randomized to blinded treatment with heparin-saline placebo catheter lock therapy.
  Interventions: Drug: heparin-saline placebo

INTERVENTIONS:
Drug: ethanol — 70% ethanol catheter lock therapy
  Other Names: 70% ethanol
  Arms: Treatment
Drug: heparin-saline placebo — heparin-saline placebo catheter lock therapy
  Other Names: heparin-saline
  Arms: Control

SUMMARY:
Use of long-term central venous access devices (including tunneled lines and ports) can be associated with development of bloodstream infection caused by build-up of bacteria or fungus on the inside of the device, called central line associated bloodstream infection (CLABSI). This infection generally requires hospital admission and antibiotic therapy. This treatment usually helps eradicate the infection but sometimes it is not possible to clear or it comes back after treatment. Also, once someone has had one line infection the chance of getting another one is higher. This study will test whether treatment and secondary prophylaxis of CLABSI with ethanol lock therapy (ELT) can significantly reduce the risk of treatment failure (comprising failure to clear initial infection, relapse or reinfection) in children and adolescents treated for cancer or hematologic disorders or undergoing hematopoietic stem cell transplantation (HSCT). ELT involves injecting a solution of ethanol and water into the line or port, allowing it to dwell for 2 hours, and then withdrawing the solution.

DETAILED DESCRIPTION:
Eligible patients with CLABSI will be enrolled within 96 hours of collection of positive blood culture and randomized to blinded treatment with 70% ethanol or heparin-saline placebo catheter lock therapy.

After enrollment, all subjects will receive catheter lock therapy for a 5 day Treatment Phase, followed by a 24 week Prophylaxis Phase. Participants in the active treatment arm will receive 70% ethanol locks and those in the placebo arm will receive heparin-saline placebo locks in identical fashion.

In addition to the study intervention, participants in both arms will receive standard systemic antibiotic therapy according to the preference of the ward clinician.

The intervention will continue for 24 weeks unless off-therapy criteria are met or the catheter is removed.

After the intervention is discontinued, participants will be monitored for 90 days, or 30 days after line removal, whichever is shorter. If the intervention is discontinued prior to 24 weeks due to adverse event or physician request, participants will be monitored for the remainder of the 24 week period.

Primary Objective:

* To compare the proportion of therapeutic failures in children and adolescents with CLABSI during treatment with standard care plus Ethanol Lock Therapy (ELT) versus standard care alone.

Secondary Objectives:

* To estimate and compare the cumulative incidence of CLABSI treatment failure, relapse or reinfection in children and adolescents receiving ELT plus standard care versus those receiving standard care alone.
* To estimate the risk of central venous access device (CVAD) occlusion associated with the use of ELT plus standard care, compared with standard care alone, in children and adolescents.
* To estimate the risk of adverse events possibly attributable to ELT associated with the use of ELT plus standard care, compared with standard care alone, in children and adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Subjects ≥6 months to < 25 years of age who are ≥5kg
* New diagnosis (within 96 hours of collection of first positive blood culture) of CLABSI (participants with previous CLABSI will be eligible if not previously enrolled in the study)
* Silicone CVAD in situ (ports, Hickman and Broviac lines will all be eligible)
* Treating clinician plans to attempt salvage of CVAD
* Participant is receiving treatment for cancer or any hematologic disorder or is receiving hematopoietic stem cell transplantation (HSCT) at a participating institution.

Exclusion Criteria:

* Allergy to ethanol or components of placebo lock
* Concomitant use of metronidazole, disulfiram or trabectedin
* Plan to remove CVAD within 6 days
* Continuous use of all lumens of CVAD leading to anticipated inability to lock each lumen for at least 2 hours per day
* Known CVAD obstruction
* Subjects who are capable of becoming pregnant will require an negative pregnancy test before entry to study
* Use of ELT in the preceding 2 weeks
* Expected survival <6 days
* Proven alternative source of bloodstream infection (BSI), or clinical evidence of CVAD track or port-pocket infection
* Multiple long-term CVADs in situ

Ages: 6 Months to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 95 (Actual)
Dates: Start 2011-12-29 (Actual); Primary Completion 2016-11-11 (Actual); Study Completion 2016-11-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Wolf, MBBS, BA, Principal Investigator — St. Jude Children's Research Hospital
Locations (2):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States
- Royal Children's Hospital Melbourne, Parkville, Victoria, Australia

REFERENCES:
- [Derived] Wolf J, Connell TG, Allison KJ, Tang L, Richardson J, Branum K, Borello E, Rubnitz JE, Gaur AH, Hakim H, Su Y, Federico SM, Mechinaud F, Hayden RT, Monagle P, Worth LJ, Curtis N, Flynn PM. Treatment and secondary prophylaxis with ethanol lock therapy for central line-associated bloodstream infection in paediatric cancer: a randomised, double-blind, controlled trial. Lancet Infect Dis. 2018 Aug;18(8):854-863. doi: 10.1016/S1473-3099(18)30224-X. Epub 2018 Jun 5. PMID 29884572
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants meeting eligibility criteria were enrolled between December 2011 and August 2016. They were randomized to receive catheter lock therapy using either 70% ethanol or heparin-saline (placebo). Randomization was blinded to the participant, their care provider, the investigator, and the outcomes assessor.
Groups:
- Treatment (Ethanol): Eligible patients with CLABSI will be enrolled within 96 hours of collection of positive blood culture and randomized to blinded treatment with 70% ethanol catheter lock therapy.
  ethanol: 70% ethanol catheter lock therapy
- Control (Placebo): Eligible patients with CLABSI will be enrolled within 96 hours of collection of positive blood culture and randomized to blinded treatment with heparin-saline placebo catheter lock therapy.
  heparin-saline placebo: heparin-saline placebo catheter lock therapy
Period: Overall Study
Arm/Group | Treatment (Ethanol) | Control (Placebo)
Started | 49 | 46
Completed | 48 | 46
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment (Ethanol) | Control (Placebo) | Total
Number analyzed (Participants) | 48 | 46 | 94
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.8 (6.3) | 8.3 (6.7) | 8.6 (6.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 21 | 35
  Male | 34 | 25 | 59
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 8 | 16
  Not Hispanic or Latino | 35 | 36 | 71
  Unknown or Not Reported | 5 | 2 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 6 | 12 | 18
  White | 31 | 30 | 61
  More than one race | 4 | 1 | 5
  Unknown or Not Reported | 3 | 2 | 5
Region of Enrollment [Number; unit: participants]
  United States | 42 | 45 | 87
  Australia | 6 | 1 | 7

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Therapeutic Failures (Early or Late Failure) in Children and Adolescents With CLABSI Receiving Standard Care Plus Ethanol Lock Therapy (ELT) vs. Standard Care Alone
Description: Therapeutic failure was a pre-defined composite outcome comprising either 'early failure': central line removal, death, persistent positive blood cultures for >72 hours, development of new CLABSI, or initiation of other ALT) during the 5 day treatment phase, or 'late failure': relapse (new CLABSI with an identical organism), or reinfection (new CLABSI with a different organism) during the 24 week prophylaxis phase. The percentage of evaluable participants with therapeutic failure is reported.
Time Frame: Up to 25 weeks after the start of treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Treatment (Ethanol) | Control (Placebo)
Number analyzed (Participants) | 48 | 46
percentage of participants | 43.8 | 43.5

2. Secondary Outcome: Cumulative Incidence of Therapeutic Failure in Participants Receiving Standard Care Plus ELT vs. Standard Care Alone
Description: Therapeutic failure was a pre-defined composite outcome comprising either 'early failure': central line removal, death, persistent positive blood cultures for >72 hours, development of new CLABSI, or initiation of other ALT) during the 5 day treatment phase, or 'late failure': relapse (new CLABSI with an identical organism), or reinfection (new CLABSI with a different organism) during the 24 week prophylaxis phase. The cumulative incidence of therapeutic failure is reported.
Time Frame: Up to 25 weeks after the start of treatment
Measure: Number; unit: percentage of participants
Arm/Group | Treatment (Ethanol) | Control (Placebo)
Number analyzed (Participants) | 48 | 46
percentage of participants | 44.0 | 43.9

3. Secondary Outcome: Cumulative Incidence of Relapse in Participants Receiving Standard Care Plus ELT vs. Standard Care Alone
Description: Relapse was defined as new CLABSI with an identical organism occurring during the 24 week prophylaxis phase. The percentage of evaluable participants with relapse is reported.
Time Frame: Up to 25 weeks after the start of treatment
Measure: Number; unit: percentage of participants
Arm/Group | Treatment (Ethanol) | Control (Placebo)
Number analyzed (Participants) | 48 | 46
percentage of participants | 6.3 | 8.7

4. Secondary Outcome: Cumulative Incidence of Reinfection in Participants Receiving Standard Care Plus ELT vs. Standard Care Alone
Description: Reinfection was defined as new CLABSI with a different organism occurring during the 24 week prophylaxis phase. The percentage of evaluable participants with reinfection is reported.
Time Frame: Up to 25 weeks after the start of treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Treatment (Ethanol) | Control (Placebo)
Number analyzed (Participants) | 48 | 46
percentage of participants | 27.3 | 24.4

5. Secondary Outcome: Rate of Central Venous Access Device (CVAD) Occlusion Events in Participants Receiving Standard Care Plus ELT vs. Standard Care Alone
Description: Occlusion was defined as central line occlusion or dysfunction requiring thrombolytic therapy. The percentage of evaluable participants requiring thrombolytic therapy for central line occlusion is reported.
Time Frame: Up to 26 weeks after the start of treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Treatment (Ethanol) | Control (Placebo)
Number analyzed (Participants) | 48 | 46
percentage of participants | 58.3 | 32.6

6. Secondary Outcome: Adverse Events in Participants Receiving Standard Care Plus ELT vs. Standard Care Alone
Description: Adverse events attributable to lock therapy or related to the central venous access device (CVAD) were elicited from direct questioning at study visits and from the medical record. The percentage of evaluable participants with any potentially attributable adverse effect is reported.
Time Frame: Up to 37.5 weeks after the start of treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Treatment (Ethanol) | Control (Placebo)
Number analyzed (Participants) | 48 | 46
percentage of participants | 60.4 | 39.1

ADVERSE EVENTS:
Time Frame: Adverse events were collected from on study date through through off study date (up to 263 days).
Description: Adverse events attributable to lock therapy or related to the central venous access device (CVAD) were elicited from direct questioning at study visits and from the medical record.
Arm/Group | Treatment (Ethanol) | Control (Placebo)
All-Cause Mortality (participants affected / at risk) | 3/48 | 4/46
Serious Adverse Events (participants affected / at risk) | 6/48 | 5/46
Other Adverse Events (participants affected / at risk) | 4/48 | 0/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Ethanol) (N=48) | Control (Placebo) (N=46)
Line fracture or split (Product Issues) | 6 (6) | 4 (4)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Ethanol) (N=48) | Control (Placebo) (N=46)
Chest pain (infusional) (General disorders) | 4 (4) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes